CLINICAL TRIAL: NCT00790998
Title: A Single-Dose, Ivermectin-Controlled, Double-Blind, Efficacy, Safety And Tolerability Study Of Orally Administered Moxidectin In Subjects Infected With Onchocerca Volvulus
Brief Title: Study Comparing Moxidectin And Ivermectin In Subjects With Onchocerca Volvulus Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medicines Development for Global Health (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3110A1-3000; B1751006 - ONCBL60801
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2013-11

CONDITIONS: Onchocerciasis
Keywords: onchocerciasis; river blindness; onchocerca volvulus; moxidectin; ivermectin
MeSH Terms: conditions — Onchocerciasis; Onchocerciasis, Ocular | interventions — moxidectin; Ivermectin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moxidectin (Experimental): Moxidectin 8mg
  Interventions: Drug: Moxidectin
- Ivermectin (Active Comparator): Ivermectin 150 mcg/kg
  Interventions: Drug: Ivermectin

INTERVENTIONS:
Drug: Moxidectin — Single dose of moxidectin 2 mg oral tablet x 4
  Arms: Moxidectin
Drug: Ivermectin — Single dose of ivermectin 3 mg oral tablet x 2, 3 or 4
  Other Names: Ivermectin, Mectizan, Stromectol
  Arms: Ivermectin

SUMMARY:
This is a Phase 3 study comparing the efficacy, safety and tolerability of moxidectin and ivermectin in subjects infected with Onchocerca volvulus, which is the parasite that causes river blindness. Subjects participating in the study will be randomly assigned (by a 2 to1 ratio) to receive one orally-administered dose of either moxidectin or ivermectin.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with Onchocerca volvulus infection

Exclusion Criteria:

* Pregnant or breast feeding women; coincidental loiasis

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1497 (Actual)
Dates: Start 2009-04; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
skin microfilaria density (mf/mg) | 12 months

SECONDARY OUTCOMES:
skin microfilaria density (mf/mg) | 1 month
skin microfilaria density (mf/mg) | 6 months
skin microfilaria density (mf/mg) | 18 months
skin microfilaria reduction from baseline | 1 month
skin microfilaria reduction from baseline | 6 months
skin microfilaria reduction from baseline | 12 months
skin microfilaria reduction from baseline | 18 months
proportion of subjects with undetectable levels of skin microfilaria | 1 month
proportion of subjects with undetectable levels of skin microfilaria | 6 months
proportion of subjects with undetectable levels of skin microfilaria | 12 months
proportion of subjects with undetectable levels of skin microfilaria | 18 months
percent reduction in microfilaria levels in the anterior chamber of the eye | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Special Programme for Research and Training in Tropical Diseases (TDR), Study Director — World Health Organization
Locations (4):
- Democratic Republic of the Congo (2):
  - Centre de Recherche Clinique de Butembo - Université Catholique du Graben, Butembo
  - Centre de Recherche en Maladies Tropicales de l'Ituri, Rethy
- Onchocerciasis Chemotherapy Research Center, Hohoe, Ghana
- Liberian Institute for Biomedical Research Clinical Research Center, Bolahun, Lofa County, Liberia

REFERENCES:
- [Result] Opoku NO, Bakajika DK, Kanza EM, Howard H, Mambandu GL, Nyathirombo A, Nigo MM, Kasonia K, Masembe SL, Mumbere M, Kataliko K, Larbelee JP, Kpawor M, Bolay KM, Bolay F, Asare S, Attah SK, Olipoh G, Vaillant M, Halleux CM, Kuesel AC. Single dose moxidectin versus ivermectin for Onchocerca volvulus infection in Ghana, Liberia, and the Democratic Republic of the Congo: a randomised, controlled, double-blind phase 3 trial. Lancet. 2018 Oct 6;392(10154):1207-1216. doi: 10.1016/S0140-6736(17)32844-1. Epub 2018 Jan 18. PMID 29361335
- [Derived] Bakajika D, Kanza EM, Opoku NO, Howard HM, Mambandu GL, Nyathirombo A, Nigo MM, Kennedy KK, Masembe SL, Mumbere M, Kataliko K, Bolay KM, Attah SK, Olipoh G, Asare S, Vaillant M, Halleux CM, Kuesel AC. Effect of a single dose of 8 mg moxidectin or 150 mug/kg ivermectin on O. volvulus skin microfilariae in a randomized trial: Differences between areas in the Democratic Republic of the Congo, Liberia and Ghana and impact of intensity of infection. PLoS Negl Trop Dis. 2022 Apr 27;16(4):e0010079. doi: 10.1371/journal.pntd.0010079. eCollection 2022 Apr. PMID 35476631
- See also: Single dose moxidectin versus ivermectin for Onchocerca volvulus infection in Ghana, Liberia, and the Democratic Republic of the Congo: a randomised, controlled, double-blind phase 3 trial — http://dx.doi.org/10.1016/S0140-6736(17)32844-1